CLINICAL TRIAL: NCT04478279
Title: A Phase 1-2 Dose-escalation and Expansion Study of ST101 in Patients With Advanced Unresectable and Metastatic Solid Tumors
Brief Title: A Phase 1-2 Study of ST101 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sapience Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST101-101
Record Dates: First submitted 2020-07-02; First posted 2020-07-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma; Melanoma Stage IV; Breast Cancer; Prostate Cancer; Glioblastoma Multiforme; GBM; Brain Cancer; Metastatic Breast Cancer; Metastatic Melanoma; Metastatic Prostate Cancer; Melanoma Recurrent; Prostate Cancer Metastatic; Recurrent Glioblastoma; Newly Diagnosed Glioblastoma
MeSH Terms: conditions — Glioblastoma; Melanoma; Breast Neoplasms; Prostatic Neoplasms; Brain Neoplasms | interventions — Temozolomide; Radiation

STUDY DESIGN:
Intervention Model Description: The study consists of two phases: a phase 1 dose escalation/regimen exploration phase and a phase 2 expansion phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Escalation (Experimental): This cohort only patients diagnosed with locally advanced or metastatic melanoma, carcinoma or sarcoma of any tumor type who are refractory or intolerant to all available therapies. ST101 will be administered intravenously (IV), initially once per week.
  Interventions: Drug: ST101
- Dose Expansion HR+ Breast (Experimental): This cohort must have progressed after 1-2 hormone based therapies. The starting dose of ST101 for Expansion will be derived from the maximum tolerated dose (MTD)/recommended dose for expansion (RDE) and the best dosing schedule determined during Dose Escalation.
  Interventions: Drug: ST101
- Dose Expansion Melanoma (Experimental): This cohort must have Melanoma that has progressed after/or on treatment with an immune checkpoint inhibitor (CPI) and have received 1-2 prior lines of therapy for their advanced/metastatic disease. The starting dose of ST101 for Expansion will be derived from the maximum tolerated dose (MTD)/recommended dose for expansion (RDE) and the best dosing schedule determined during Dose Escalation.
  Interventions: Drug: ST101
- Dose Expansion GBM (Experimental): Primary (de novo) GBM that has recurred or progressed (per modified RANO criteria) after 1 standard treatment regimen. Standard therapy is defined as maximal surgical resection, radiotherapy, and concomitant temozolomide with radiotherapy or adjuvant chemotherapy with temozolomide. The starting dose of ST101 for Expansion will be derived from the maximum tolerated dose (MTD)/recommended dose for expansion (RDE) and the best dosing schedule determined during Dose Escalation.
  Interventions: Drug: ST101
- Dose Expansion CRPC (Experimental): CRPC that has progressed after previous treatment with taxanes, abiraterone and enzalutamide/apalutamide. The starting dose of ST101 for Expansion will be derived from the maximum tolerated dose (MTD)/recommended dose for expansion (RDE) and the best dosing schedule determined during Dose Escalation.
  Interventions: Drug: ST101
- Dose Expansion Recurrent Glioblastoma (Experimental): Recurrent GBM patients must have completed radiation at least 3 months prior to minimize the inclusion of patients with pseudoprogression. Recurrent GBM patients must have unequivocal radiographic evidence of tumor progression by contrast-enhanced magnetic resonance imaging (MRI) scan within 21 days prior to registration. Patients must be able to delay surgery for 2 - 4 weeks per investigator decision
  Interventions: Drug: ST101
- Newly Diagnosed Glioblastoma (Experimental): Newly diagnosed patients with a suboptimal resection or biopsy must be candidates for another surgical resection as determined by neurosurgical evaluation or multidisciplinary team based on the current standard of care that suggests that maximal safe resection is beneficial. Recurrent GBM patients must be candidates for tumor resection
  Interventions: Drug: ST101; Drug: Temozolomide; Radiation: Radiation

INTERVENTIONS:
Drug: ST101 — ST101 will be administered intravenously (IV), initially once per week with a flat dose on the schedule described for each study arm
Drug: Temozolomide — Temozolomide
  Arms: Newly Diagnosed Glioblastoma
Radiation: Radiation — Radiation
  Arms: Newly Diagnosed Glioblastoma

SUMMARY:
This is an open-label, two-part, phase 1-2 dose-finding study designed to determine the safety, tolerability, PK, PD, and proof-of-concept efficacy of ST101 administered IV in patients with advanced solid tumors. The study consists of two phases: a phase 1 dose escalation/regimen exploration phase and a phase 2 expansion phase.

DETAILED DESCRIPTION:
Dose escalation / regimen exploration phase During the dose escalation/regimen exploration phase, only patients diagnosed with locally advanced or metastatic melanoma, carcinoma or sarcoma of any tumor type who are refractory or intolerant to all available therapies that would impact survival will be enrolled.

ST101 will be administered intravenously (IV), initially once per week. The dose escalation cohorts will be recruited using a standard 3+3 design. At each new dosing cohort, there will be a 1-week observation period after dosing the first patient in order to assess safety prior to dosing the remainder of the patients in that cohort. The dose cohorts will be 0.5, 1, 2, 4, 8 and 16 mg/kg with once weekly (QW) dosing in all cohorts except for the highest dose level which will be dosed every other week (Q2W).

The expansion phase consists of 4 specific tumor-type cohorts, which each follow the same Simon 2-stage design. Fifteen (15) patients will be enrolled in each cohort and treated with the ST101 RP2D. If one or more responses is observed that cohort will be expanded to a total of 30 patients to further assess efficacy.

Responses will be graded using response evaluation criteria in solid tumors (RECIST) 1.1 (Eisenhauer 2009) for hormonal receptor positive (HRpos) locally advanced/metastatic breast cancer (LA/MBC) and melanoma, modified response assessment in neuro-oncology (RANO) (Ellingson 2017) for GBM and prostate cancer clinical trials working group 3 (PCWG3) (Scher 2016) for castration-resistant prostate cancer (CRPC).During the expansion phase, only patients diagnosed with the following tumor types will be allowed into this phase of the study:

* HRpos LA/MBC that has progressed after prior 1-2 hormone-based therapies. Previous treatment with cyclin-dependent kinase 4/6 (CDK4/6) inhibitor, mammalian target of rapamycin (mTOR) inhibitor or chemotherapy is allowed as monotherapy or in combination.
* Melanoma that has progressed after/or on treatment with an immune checkpoint inhibitor (CPI) and have received 1-2 prior lines of therapy for their advanced/metastatic disease. Patients that have BRAF mutated disease should also have received one line of appropriate targeted therapy.
* Primary (de novo) GBM that has recurred or progressed (per modified RANO criteria) after 1 standard treatment regimen. Standard therapy is defined as maximal surgical resection, radiotherapy, and concomitant temozolomide with radiotherapy or adjuvant chemotherapy with temozolomide. Patients that undergo tumor treating fields as an adjuvant to first line therapy are allowed.
* CRPC that has progressed after previous treatment with taxanes, abiraterone and enzalutamide/apalutamide.

The tumor types in the expansion phase may change based on emerging data from the dose escalation phase of this study. Additional mini cohorts of 10 patients may be added to the expansion phase based on efficacy signals during the dose escalation phase.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Able and willing to sign informed consent form (ICF) and comply with the protocol and the restrictions and assessments therein.
  2. Male or female ≥18 years of age.
  3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
  4. Must have a locally advanced or metastatic inoperable tumor as follows:

     1. For the dose escalation/regimen exploration phase: melanoma, carcinoma, or sarcoma
     2. For the expansion phase: HR positive LA/MBC, melanoma, GBM, CRPC
  5. Agrees to provide a newly obtained biopsy of an accessible lesion (if they can be biopsied based on the investigator's assessment) prior to the start of study treatment, and to repeat biopsy once during study treatment. Tissue obtained for the biopsy must not be previously irradiated (unless progressing following irradiation), but a new or progressing lesion in the radiation field is acceptable. Archived biopsies are acceptable for GBM patients.
  6. In the investigator's opinion, the patient may not derive clinical benefit from, or is ineligible for, a particular form of standard therapy on medical grounds, or the patient failed or did not tolerate one or more of other anti-cancer therapies:

     a. For the dose escalation/regimen exploration phase up to 3 previous lines of systemic anticancer therapies are allowed. Since this is a FIH study, it's important that patients are not refractory to therapeutic intervention due to multiple lines of prior therapies.

     a. For the expansion phase: i. HRpos LA/MBC must have progressed after prior 1-2 hormone-based therapies. Previous treatment with cyclin-dependent kinase 4/6 (CDK4/6) inhibitor, mammalian target of rapamycin (mTOR) inhibitor or chemotherapy is allowed as monotherapy or in combination ii. Melanoma that has progressed after or on treatment with a CPI and have received 1-2 prior lines of therapy for their advanced/metastatic disease. Patients that have BRAF mutated disease should also have received one line of appropriate targeted therapy iii. Primary (de novo) GBM that has recurred or progressed (per modified RANO criteria) after 1 standard treatment regimen (surgery, radiotherapy, and temozolomide therapy). Patients that undergo tumor treating fields as an adjuvant to first line therapy are allowed.

     iv. CRPC that has progressed after previous treatment with taxanes, abiraterone and enzalutamide/apalutamide or that are intolerant to these treatments.
  7. Evaluable disease per RECIST 1.1, modified RANO or PCWG3 with at least one target lesion
  8. Disease that progressed on, or is non-responsive to, the previous line of therapy per RECIST 1.1, modified RANO or PCWG3.
  9. If not menopausal or surgically sterile, willing to practice at least one of the following highly effective methods of birth control for at least a (partner's) menstrual cycle before and for four months after ST101 administration: (1) total abstinence from sexual intercourse with a member of the opposite sex; (2) sexual intercourse with vasectomized male/sterilized female partner; (3) combined (estrogen and progestogen containing) or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, parenteral, transvaginal or transdermal) for at least 3 consecutive months prior to investigational product administration; (4) other acceptable forms of birth control (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicide or cream); (5) use of an intrauterine contraceptive device.
  10. All previous anti-cancer therapy-related adverse events should have resolved to grade 1 or baseline value with the exception of alopecia. Levothyroxine is allowed for patients that previously received a CPI and experienced thyroid dysfunction.

      Exclusion Criteria

  <!-- -->

  1. Use of small molecule or tyrosine kinase inhibitor within 2 weeks or 5 half-lives (whichever is shorter) prior to the first dose of study drug; chemotherapy, investigational drug or biological cancer therapy within 3 weeks prior to the first dose of study therapy; nitrosourea or radioisotope within 6 weeks prior to first dose.
  2. Known hypersensitivity to ST101 or any of its excipients.
  3. Baseline corrected interval between q and t wave on electrocardiogram (ECG) (QTc) > 480 msec using Fredericia's formula.
  4. Symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
  5. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging brain metastases, and are off steroids for at least 14 days prior to first dose of study drug. This criterion does not apply to patients on the GBM cohort.
  6. Presence of any other active malignancy requiring systemic therapy other than the disease under study.
  7. Active infection with human immunodeficiency virus (HIV) and CD4+ T-cell count <350/μL. Patients not on established ART for at least four weeks and having a detectable HIV viral load. Testing is not required for eligibility.
  8. Active infection with hepatitis B or hepatitis C, defined by a detectable viral load. Testing is not required for eligibility.
  9. Active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Vitiligo or resolved childhood asthma/atopy are exceptions to this rule. Patients requiring intermittent use of bronchodilators or topical steroids would not be excluded from the study. Patients with hypothyroidism that is stable on hormone replacement or controlled type 1 diabetes will not be excluded from the study.
  10. Use of systemic corticosteroids to treat inflammatory or autoimmune symptoms within 15 days or other immunosuppressive drugs within 30 days prior to the start of the study. Inhaled and topical corticosteroids are permitted. Up to 10 mg/day prednisone or equivalent is permitted as replacement therapy for adrenal insufficiency only.
  11. Active infection requiring systemic therapy.
  12. Active immune thrombocytopenic purpura or other chronic thrombocytopenic condition.
  13. Therapeutic anticoagulation that cannot be interrupted for a biopsy or had a thromboembolic event within the last 6 months.
  14. History or clinical evidence of any surgical or medical condition which the investigator judges as likely to interfere with the results of the study or pose an additional risk in participating, or makes the patient unlikely to comply with the study related visits and assessments particularly any pre-existing condition that would put the patient at additional risk should they experience an infusion-related reaction, e.g., rapidly progressive or uncontrolled disease involving a major organ system - vascular, cardiac, pulmonary, gastrointestinal, gynecologic, hematologic, neurologic, neoplastic, renal, endocrine, or an immunodeficiency
  15. Unable to comply with the visits and requirements of the protocol due to psychiatric condition or substance abuse. Pregnant or breastfeeding or planning to conceive or father children within the projected duration of the study.
  16. Exclusion Criteria for GBM Cohort:

      a) Any prior therapy for GBM other than that which is considered SOC for primary GBM, including but not limited to the following: i. more than one line of adjuvant temozolomide ii. prior treatment with another investigational drug iii. prior treatment with bevacizumab (Avastin) or other vascular-endothelial growth factor (VEGF) inhibitors or VEGF-receptor signaling inhibitors iv. prior treatment with nitrosoureas v. prior therapy that included interstitial brachytherapy or Gliadel® Wafers (carmustine implants) b) secondary GBM (i.e., GBM that progressed from low-grade diffuse astrocytoma or AA) c) tumor with a clinically significant mass effect (>5 mm midline shift) while on a stable corticosteroid dose d) prednisone or equivalent dose of >10mg per day e) known history of allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 20 months
  Number of Participants with a Dose-Limiting Toxicity (DLT)
Adverse Events | 20 months
  Number of Participants with at Least One Adverse Event, Severity Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)

SECONDARY OUTCOMES:
Area Under the Curve (AUC) | 30 Months
  Area under the plasma concentration time curve of ST101
Cmax | 20 months
  Peak plasma concentration of ST101
Terminal Half-Life (t1/2) | 20 months
  Elimination half-life of ST101
Overall Response | 20 months
  Escalation and Expansion Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
DCR | 20 Months
  Expansion: Disease Control Rate, Assessed According to RECIST v1.1
Duration of Response | 20 months
  Expansion: Duration of Response, Assessed According to RECIST v1.1
PFS | 20 months
  Expansion: Progression Free Survival, Assessed According to RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Abi Vainstein-Haras, MD, Study Chair — CMO
Locations (11):
- United States (7):
  - University of California, San Francisco, San Francisco, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Northwestern Medicine Cancer Centers, Warrenville, Illinois
  - START Midwest, Grand Rapids, Michigan
  - Columbia University, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
- United Kingdom (4):
  - Edinburgh Cancer Centre, Edinburgh
  - The Beaston West of Scotland Cancer Centre, Glasgow
  - University of Leeds, Leeds
  - Sarah Cannon Research Institute UK, London

IPD SHARING:
Plan to Share IPD: No